CLINICAL TRIAL: NCT00221442
Title: Zonegran in the Treatment of Binge Eating Disorder Associated With Obesity: A Single Center, Double-Blind, Placebo-controlled, Flexible-Dose Study in Outpatients
Brief Title: Zonegran in the Treatment of Binge Eating Disorder Associated With Obesity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Collaborators: Eisai Inc. (Industry); University of Cincinnati (Other)
Responsible Party: Susan L .McElroy, MD / Professor, Lindner Center of HOPE
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 51-345-740
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Binge Eating Disorder Associated With Obesity
Keywords: Adults; Binge eating disorder; Blood draw; E.Coli enterprotoxin; Eating disorders; Electrocardiogram; Females; Males; Physical exam; Psychiatric evaluation; Questionnaire
MeSH Terms: conditions — Binge-Eating Disorder; Feeding and Eating Disorders | interventions — Zonisamide; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- zonisamide (Active Comparator): zonegran (zonisamide)
  Interventions: Drug: Zonegran
- Sugar pill (Placebo Comparator): fake pill
  Interventions: Drug: sugar pill

INTERVENTIONS:
Drug: Zonegran — zonegran (zonisamide)
  Arms: zonisamide
Drug: sugar pill — fake pill
  Arms: Sugar pill

SUMMARY:
The specific aim of this study is to examine the efficacy and safety of zonisamide compared with placebo in outpatients with binge eating disorder associated with obesity.

DETAILED DESCRIPTION:
Binge eating disorder (BED) is characterized by recurrent, uncontrollable, and distressing episodes of excessive food consumption (binge eating) without compensatory weight loss behaviors.1,2 Its prevalence in the general population of the United States is conservatively estimated to be 1.5% to 2%,1-6 making it more common than anorexia nervosa and bulimia nervosa combined. BED is associated with being overweight and obesity.1-7 Approximately 8% to 30% of those seeking standard weight loss treatments, 1-4 up to 50% of those seeking bariatric surgery,8,9 and 70% of those participating in Overeaters Annonymous3 are estimated to have BED.

Zonisamide is a structurally and pharmacologically novel antiepileptic drug - a sulfamate-substituted monosaccharide - with proven anticonvulsant efficacy when used adjunctively in refractory partial epilepsy.10-12 Mechanisms hypothesized to account for zonisamide's antiepileptic properties include antagonism of voltage-gated sodium and T-type calcium channels, blockade of potassium-evoked glutamate release, modulation of central dopaminergic and serotonergic function, and carbonic anhydrase inhibition.10-16 Several lines of evidence suggest that zonisamide might be a useful treatment for BED. First, like the anticonvulsant topiramate,17-19 zonisamide has been associated with anorexia and weight loss in clinical trials in epilepsy patients10,11,20 and in patients with obesity.20 Topiramate has also been shown to reduce binge eating and weight in patients with binge eating disorder associated with obesity. 21 Although zonisamide and topiramate have distinct pharmacologic profiles, both drugs share several pharmacologic actions. These include sodium channel blockade, carbonic anhydrase inhibition, and reduction of glutamate neurotransmission. 10,11,13,16,17 Regarding the latter property, animal studies have shown that stimulation of the lateral hypothalamus by glutamate and glutamate agonists causes an intense, rapid, dose-dependent increase in food intake,22 whereas glutamate antagonism of the nucleus tractus solitarius reduces food intake.23 Second, unlike topiramate, zonisamide also modulates the function of serotonin and dopamine14, 15 --two neurotransmitters involved in the regulation of feeding behavior24 and the mechanisms of some medications with efficacy in either binge eating (SSRIs, d-fenfluramine) 25-29 or obesity (sibutramine, stimulants).30 Third, a broad range of antidepressants have been reported to reduce binge eating in both bulimia nervosa31 and binge eating disorder25-28,32 and preliminary observations suggest zonisamide may have thymoleptic properties.33,34 Fourth, in an open-label trial of zonisamide in 15 patients with BED conducted by our group, zonisamide was effective in reducing binge eating frequency, severity of illness, and weight (S.L. McElroy, J Clin Psychiatry, under review).35 We therefore propose to conduct a double-blind, placebo-controlled, randomized, parallel group, 16-week study of zonisamide in 60 outpatients with binge eating disorder and obesity.

ELIGIBILITY:
Inclusion Criteria:

Patients will meet DSM-IV criteria for BED for at least the last 6 months. These criteria are as follows:

* Recurrent episodes of binge eating. An episode of binge eating is characterized by both of the following: (1) eating, in discrete period of time (eg, within any two hour period), an amount of food that is definitely larger than most people would eat in a similar period of time under similar circumstances and (2) a sense of lack of control over eating during the episode (eg, a feeling that one cannot stop eating or control what or how much one is eating)
* The binge eating episodes are associated with at least three of the following:

  * Eating much more rapidly than normal
  * Eating until uncomfortably full
  * Eating large amounts of food when not feeling physically hungry
  * Eating alone because of being embarrassed by how much one is eating
  * Feeling disgusted with oneself, depressed, or feeling very guilty after overeating
* Marked distress regarding binge eating.
* The binge eating occurs, on average, at least two days a week for six months.
* Does not occur exclusively during the course of bulimia nervosa and anorexia nervosa.
* Obesity as defined by body mass index > 30 kg/m2.
* Men or women, between the ages of 18 and 65. The patient population is expected to be predominantly made up of women based on previous research.

Exclusion Criteria:

* Have current body mass index < 30kg/m2.
* Women who are pregnant or lactating and women of childbearing potential who are not taking adequate contraceptive measures. If there is a possibility a female subject might be pregnant, a pregnancy test will be performed. (All women of childbearing potential will have a negative pregnancy test before entering the study.)
* Subjects who are displaying clinically significant suicidality or homicidality.
* Subjects who are displaying a current clinically unstable depressive disorder (e.g., HAM-D > 21).
* A current or recent (within 6 months of the start of study medication) DSM-IV diagnosis of substance abuse or dependence.
* A lifetime history of a DSM-IV bipolar disorder or dementia.
* History of a personality disorder (eg, schizotypal, borderline, or antisocial) which might interfere with assessment or compliance with study procedures.
* Clinically unstable medical disease, including cardiovascular, hepatic, renal, gastrointestinal, pulmonary, metabolic, endocrine or other systemic disease which could interfere with diagnosis, assessment, or treatment of binge eating disorder. Patients should be biochemically euthyroid prior to entering the study.
* History of seizures, including febrile seizures in childhood
* History of clinically significant nephrolithiasis.
* Subjects requiring treatment with any drug which might interact adversely with or obscure the action of the study medication (e.g. stimulants, sympathomimetics, antidepressants, carbonic anhydrase inhibitors, anti-obesity drugs).
* Subjects who have received psychoactive medication (other than zaleplon [Sonata] or zolpidem [Ambien] -- as needed for restlessness/insomnia) within one week prior to randomization.
* Subjects who have begun and/or are receiving formal psychotherapy (cognitive behavioral therapy, interpersonal therapy, or dietary behavioral therapy) for BED or weight loss within the past 3 months.
* Subjects previously enrolled in this study or have previously been treated with zonisamide.
* Subjects who have received an experimental drug or used an experimental device within 30 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
frequency of binge eating episodes | per protocol

CONTACTS AND LOCATIONS:
Overall Officials: Susan L McElroy, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Result] McElroy SL, Kotwal R, Guerdjikova AI, Welge JA, Nelson EB, Lake KA, D'Alessio DA, Keck PE, Hudson JI. Zonisamide in the treatment of binge eating disorder with obesity: a randomized controlled trial. J Clin Psychiatry. 2006 Dec;67(12):1897-906. doi: 10.4088/jcp.v67n1209. PMID 17194267